CLINICAL TRIAL: NCT01011582
Title: Human Subjects Registry of Characteristics and Outcomes of Intensive Care Unit Patients Admitted With Novel H1N1 Influenza or Seasonal Influenza
Brief Title: Characteristics and Outcomes of Intensive Care Unit Patients Admitted With Novel H1N1 Influenza or Seasonal Influenza
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: VCU IRB HM12562
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: H1N1 Influenza; Seasonal Influenza
Keywords: To evaluate biomarkers that cause critical illness in patients with novel H1N1 influenza and with seasonal influenza.
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimens and sputum specimens will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Novel H1N1 influenza
- Seasonal influenza

SUMMARY:
The purpose of this research study is to collect information on problems that patients with the novel H1N1 influenza and/or the seasonal influenza experience. Novel H1N1 flu is also called the swine flu. Seasonal influenza is also called the regular flu. The purpose of this study is to collect information from patients who are infected with either the novel H1N1 or the seasonal flu and to determine what makes patients critically ill with these infections. The goal is to develop a registry that will aid investigators in determining specific markers that lead to development of severe illness in these infections.

DETAILED DESCRIPTION:
Patients admitted to the medical intensive care unit with either novel H1N1 infection or seasonal influenza infection may be eligible for participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical intensive care unit with a diagnosis of novel H1N1 influenza infection or with a diagnosis of seasonal influenza infection.

Exclusion Criteria:

* Prisoners
* Refusal of study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the medical intensive care unit at Virginia Commonwealth University Medical Center, Richmond, Virginia.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to contrast patients infected with novel H1N1 influenza to those infected with seasonal influenza. | Patients will be evaluated until May 31, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein de Wit, M.D., M.S., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Medical Center (formerly known as Medical College of Virginia), Richmond, Virginia, United States